CLINICAL TRIAL: NCT01082952
Title: Role of Eosinophils in the Proliferation of ASM Cells in Asthma
Brief Title: Role of Eosinophils in the Proliferation of Airway Smooth Muscle (ASM) Cells
Status: Completed | Type: Observational
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Saleh Zaid Al-Muhsen, Associate professor, King Saud University
Other Study IDs: effect of eosinophil on ASM
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Results first posted 2011-11-18 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2011-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Asthmatic patients
- Non asthmatic patients

SUMMARY:
Being a key player in Asthma, eosinophils constitute a potential target to interfere with the series of biological events leading to Asthma pathogenesis. In this proposal, the investigators hypothesize that the interaction between eosinophils and airway smooth muscle cells (ASM) cells plays an important role in airway remodeling. Hence the investigators will investigate the role of eosinophils in enhancing ASM cells proliferation resulting in airways remodeling. The investigators will also investigate the mechanism behind this phenomenon. This will then pave the way for medical (drug) interference at one or several sites in order to prevent one of the main potential reasons behind airway remodeling, namely eosinophil-derived ASM proliferation.

DETAILED DESCRIPTION:
Rational and hypothesis Asthma is a chronic inflammatory disorder of the lung airways that is associated with airway remodeling and hyperresponsiveness (AHR). Its is well documented that the smooth muscle mass in asthmatic airways is increased due to hypertrophy and hyperplasia of the ASM cells. Moreover, eosinophils have been proposed in different studies to play a major role in airway remodeling. The association between increased eosinophil numbers and asthma severity has been well documented. Here, we hypothesized that the interaction between eosinophils and ASM cells plays an important role in airway remodeling and that eosinophils modulate the airways through enhancing ASM cell proliferation.

Objectives of the study The aim of this study is to examine the effect of eosinophils on ASM cell proliferation using eosinophils isolated from asthmatic subjects.

Specific aim 1. Effect of co-culture of ASM cells with eosinophils on ASM cell proliferation.

In this specific aim, the effect of eosinophil on ASM cell proliferation will be studied by co-culturing eosinophils isolated from asthmatic and healthy patients with ASM cells in vitro. This will be done using non-stimulated eosinophils or eosinophils activated with Interleukin-5 (IL-5)and Interleukin-3 (IL-3). ASM proliferation will be monitored by determining the levels of the proliferation marker Ki-67 expression in ASM cells.

Specific aim 2. Understanding the mechanism by which eosinophils enhance ASM proliferation.

In this specific aim, we will study the mechanism by which eosinophils enhance the proliferation of ASM cells. To study if this effect of eosinophils is done through direct contact with ASM cells, we will co-culture ASM cells with eosinophils membrane fractions. Moreover, we will examine the effect of cytokines and extracellular matrix (ECM) proteins produced by eosinophils on smooth muscle cells

ELIGIBILITY:
Asthma: Patient Selection (Inclusion Criteria)

1. Subjects with documented clinical history of asthma for a period of at least 6 months prior to study entry (and a minimum of one clinic follow-up visit since initial diagnosis)
2. Willing to provide written informed consent and in the judgment of the investigator, individuals who are able to understand the informed consent process.
3. Subjects with documented clinical history (in preceding 12 months) of airway reversibility of at least 12% based on Forced Expiratory Volume (FEV1), measured pre and post inhalation of a β-2 agonist (2 puffs of albuterol using a measured dose inhaler with spacer) OR
4. Individuals with strong history of asthma but with waning, or no current symptoms may be included in the study if their asthma was well controlled using an asthma medication. Principal investigator must verify or know the clinical history of an individual before accepting him as an asthmatic individual.
5. Able to perform Spirometry/FEV1 correctly.

Exclusion Criteria

1. Age < 5 years
2. Smoking for 20 years, 1 pack/day or more.
3. Congestive heart failure.
4. Chronic Obstructive Pulmonary Disease (COPD).
5. Chronic lung disease other than asthma and COPD.
6. Bronchiectasis.

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 12 patients per group
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2010-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saleh Al-Muhsen, MD, Study Chair — King Saud University; Rabih Halwani, PhD, Principal Investigator — King Saud University
Locations (1):
- Prince Naif center for immunological research, Riyadh, Riyadh Region, Saudi Arabia

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/17088126

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment started January 2010 and ended July 2011. Recruitment was all in King Khalid Hospital, Riyadh, Saudi Arabia
Groups:
- Asthmatic Patients: Patients were severe asthmatic with high peripheral blood eosinophil counts (>5%).
- Non Asthmatic Patients: Non asthmatic patients with high eosinophil count (>3%).
Period: Overall Study
Arm/Group | Asthmatic Patients | Non Asthmatic Patients
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asthmatic Patients | Non Asthmatic Patients | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 23 (3) | 24 (2.5) | 23.5 (2.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  Saudi Arabia | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Fold Increase in ASM Proliferation Following Incubation With Eosinophils.
Description: Airway Smooth Muscle (ASM) cell proliferation was measured 24 hrs following their co-culture with eosinophil. This was determined using Ki-67 staining and flowcytometry. The fold increase in ASM proliferation was then determined.
Time Frame: one day
Population: The number of participants for each group was determined to insure proper statistical significance when analysing the effect of isolated eosinophils on ASM cells proliferation
Measure: Mean (Standard Deviation); unit: Fold increase in ASM cell proliferation
Groups:
- Asthmatic Patients: Mild asthmatic patients with high eosinophil count (>5%)
Arm/Group | Asthmatic Patients | Non Asthmatic Patients
Number analyzed (Participants) | 6 | 6
Fold increase in ASM cell proliferation | 2 (0.2) | 2 (0.3)
Statistical Analysis 1: Comparison: Asthmatic Patients vs Non Asthmatic Patients; Test type: Superiority or Other; p < 0.05, ANOVA — The p value is calculated for the results of ASM proliferation following incubation with eosinophils isolated from patients in each group. p< 0.05 was considered significant; Proliferation data was evaluated using two-way factorial ANOVA followed by Bonferroni post hoc test

2. Secondary Outcome: Fold Increase in ASM Cells Proliferation Following Treatment With Cysteinyl Leukotrienes
Description: The effect of Eosinophil release of Cysteinyl Leukotrienes on ASM proliferation was determined using blocking agents. This was determined using Ki-67 staining and flowcytometry.
Time Frame: one day
Population: Eosinophils were collected from all the participants and used to trigger ASM proliferation.
Measure: Mean (Standard Deviation); unit: Fold increase in ASM proliferation
Arm/Group | Asthmatic Patients | Non Asthmatic Patients
Number analyzed (Participants) | 6 | 6
Fold increase in ASM proliferation | 2.3 (0.2) | 2.5 (0.1)

ADVERSE EVENTS:
Description: serious and/or other [non-serious] adverse events were not collected/assessed
Arm/Group | Asthmatic Patients | Non Asthmatic Patients
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes